CLINICAL TRIAL: NCT01132989
Title: Open-label Phase 2 Pilot Study of Lenalidomide (Revlimid) as Adjuvant Treatment for Refractory Cutaneous T Cell Lymphoma
Brief Title: Open-label Pilot Study of Lenalidomide (Revlimid) as Adjuvant Treatment for Refractory Cutaneous T Cell Lymphoma
Acronym: REvMM2009
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Florida Academic Dermatology Centers (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Francisco a Kerdel,M.D, Florida Academic Dermtology Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RevMM2009
Record Dates: First submitted 2010-05-25; First posted 2010-05-28 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2010-05

CONDITIONS: Cutaneous T Cell Lymphoma
Keywords: Patients with cutaneous T cell lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide Starting Dose Based on Renal Function at Study Entry Baseline Calculated Creatinine Clearance (by Cockcroft-Gault) Starting Lenalidomide Dose 60 ml/min 25mg daily on Days 1-21 of each 28-day cycle 30 and < 60 ml/min 10mg daily on Days 1-21 of each 28-day cycle

SUMMARY:
Patients with cutaneous T cell lymphoma experience refractory and progressive disease despite current treatment, necessitating chronic disease management. In addition, there needs to be greater emphasis on combination treatment, which correlates with increased response rate, more rapid onset of response, and decreased side effect profile compared to monotherapy. The goal for the use of Lenalidomide as an adjuvant treatment in patients with refractory cutaneous T cell lymphoma is to increase response rates, maintain a durable long-term response, relieve associated symptoms, and minimize toxic side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age (at the time of signing the informed consent).
* Able to adhere to the study visit schedule and other protocol requirements.
* Histologically confirmed mycosis fungoides or Sezary syndrome
* Stage IB to IVB disease at screening (TNMB classification, see Protocol Attachment C)
* Refractory disease after at least 2 prior therapies, which may include topicals, phototherapy, bexarotene, interferon, and/or photopheresis. Patients may be currently taking these medication and therapies may be used in combination.
* Determined to have adequate baseline organ function defined as:

Hepatic: Total bilirubin ≤ 1.5 x upper limit of normal (ULN),AST and ALT ≤ 3.0 x ULN

* Hematologic: Platelets ≥ 75 x 109/L
* Absolute neutrophil count (ANC) ≥ 1.0 x 109/L,Hemoglobin ≥ 8.0 mg/dL
* Renal: Creatinine clearance ≥ 30 ml/min (Appendix; Cockcroft-Gault formula)

  * At least 3 months since the initiation of any new CTCL treatments.
  * Stable or progressive disease despite current treatment regimen over the last 3 months.
  * All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
  * Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours prior to prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide.
  * FCBP must also agree to ongoing pregnancy testing.
  * Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.
  * A female of childbearing potential is a sexually mature woman who:

    1. has not undergone a hysterectomy or bilateral oophorectomy
    2. has not been naturally postmenopausal for at least 24 consecutive months (has had menses at any time in the preceding 24 consecutive months). See Appendix: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods.
  * Disease free of prior malignancies for ≥ 5 years, with exception of basal cell and squamous cell carcinoma of the skin, or breast or cervix in situ carcinoma.
  * Expected survival of > 6 months.
  * Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation. Patients intolerant to aspirin may use warfarin or low molecular weight heparin.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Female subjects who are pregnant, nursing, or planning pregnancy. Female subjects not using at least 2 forms of birth control during the trial, unless the subject is considered sterile (history of hysterectomy or postmenopausal with no menses for the last 24 consecutive months).
* History of deep venous thrombus (DVT) or pulmonary embolism (PE), unless currently on anticoagulation therapy (warfarin or heparin).
* Subjects receiving chemotherapeutic agents (or have received in the last 3 months), vorinostat, or methotrexate.
* Use of any other experimental drug or therapy within 28 days of baseline.
* Known hypersensitivity to thalidomide.
* History of erythema nodosum or desquamating rash while taking thalidomide or similar drugs.
* Any prior use of lenalidomide.
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine are eligible..
* Having a serious concomitant systemic disorder that could preclude the patient from benefiting or completing the study based on discretion of the investigator.
* Any condition or circumstance judged by the investigator that would render the clinical trial detrimental or otherwise unsuitable for the patient's participation.
* Neuropathy > grade 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Response rate(RR measurements are based on skin scoring using mSWAT (modified severity weighted assessment tool), Sezary cell count, and lymph node assessment. | 1 year (average)
  The primary efficacy measure is the response rate (RR) based on skin scoring using mSWAT (modified severity weighted assessment tool), Sezary cell count, and lymph node assessment. Response rate is defined as the number of responders divided by the number of treated patients. A responder is defined as any patient who exhibits a confirmed complete or partial response.
  • Patients will be treated until progressive disease is demonstrated by ≥ 25% increase of SWAT score.

SECONDARY OUTCOMES:
The assessment of patient-reported changes of pruritus during treatment | 1 year (average)
  Descriptive statistics will be calculated for pruritus relief. Both median duration of pruritus relief (for those exhibiting improvement in pruritus) and time to pruritus relief will be estimated.
The assessment of the patient-reported improvement in quality of life during treatment | 1 year (average)
  The validated DLQI patient self assessment questionnaire will be used to quantify the impact of skin disease on patients' quality of life
The assessment of the safety and tolerability of lenalidomide in the study population | 1 year (average)
  The assessments of sezary cell count ,disease status using the mSWAT tool, lymphnode evaluations and adverse event incidences( associated with study medication )will be perfomed every four weeks to assess lenalidomide safety and tolerability.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida Academic Dermatology Center, Miami, Florida, United States